CLINICAL TRIAL: NCT03812445
Title: The Effect of Probiotics on Cognition and Gut Microbiome Associated Study of Shanghai People With Acute Ischemic Stroke
Brief Title: Cognition and Gut Microbiome Associated Study of Shanghai People With Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, DIRECTOR, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cognitionstroke
Record Dates: First submitted 2019-01-03; First posted 2019-01-23 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Gastrointestinal Microbiome
Keywords: Probiotics; Gut microbiota; ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Probiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): the patients in this arm will not receive probiotics.
- Experimental (Experimental): the patients in this arm will receive probiotics blend of Bifidobacterium longum, Lactobacillus acidophilus for 3 months.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — the patients in this arm will receive probiotics blend of Bifidobacterium longum, Lactobacillus acidophilus,Bifidobacterium lactobacillus,Lactobacillus paracasei,Lactobacillus rhamnosus and Lactobacillus fermentium with does of 8*10^9 Colony-Forming Units(CFU) *2/d for 3 months.
  Arms: Experimental

SUMMARY:
The purpose of this study is to evaluate the effect of probiotics on the gut microbiome of ischemic stroke patients.

DETAILED DESCRIPTION:
This study aims to detect the impact of probiotics administration during the process of ischemic stroke treatment and recovery phase. The day of admission and 3months after stroke data will be collected and put into analysis to provide some suggestions on the probiotics use in the clinical for the stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with acute ischemic stroke on the basis of World Health Organization diagnostic criteria1.

the time from paroxysm to admission ≤2weeks.

Exclusion Criteria:

* Imaging diagnoses hemorrhagic stroke Severe depression Severe disturbance of hearing vision and reading Illiteracy Have recognitive disorder before stroke (recorded in medical records) Treated with antibiotics probiotics or prebiotics in1month before admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
change from admission on gut microbiome at 3months by genome sequencing | 3months
  change of the gut microbiome will be calculated at 3months in comparison with admission.

SECONDARY OUTCOMES:
change from admission on cognitive function at 3months by Montreal Cognitive Assessment. | 3months
  change from admission on cognitive function at 3months by Montreal Cognitive Assessment (MoCA). MoCA's score is from 0 to 30.the score is lower,the cognitive disorder is worse.
change from admission on emotion at 3months by Hamilton Depression Scale. | 3months
  change from admission on emotion at 3months by Hamilton Depression Scale（HAMD） .When HAMD's score is beyond 17,the patient is considered to have minor depression.When HAMD's score is beyond 20,the patient is considered to have medium depression. When HAMD's score is beyond 30,the patient is considered to have severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Huanlong Qin, Study Chair — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, China